CLINICAL TRIAL: NCT05238090
Title: Efficacy of a Whole Upper Limb Stretching Protocol for Lateral Epicondylitis
Brief Title: Efficacy of a Stretching Protocol for Lateral Epicondylitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cadiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPITERA
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Epicondylitis, Lateral; Elbow Tendinopathy; Epicondylitis of the Elbow; Epicondylitis
Keywords: epicondylitis; Elbow Tendinopathy; stretch; physiotherapy
MeSH Terms: conditions — Tennis Elbow; Elbow Tendinopathy

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, single-blind, multicentre, randomised study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Static stretching of the extensor carpi radialis brevis and eccentric strengthening of the wrist extensor musculature
  Interventions: Other: Static stretching of the extensor carpi radialis brevis and eccentric strengthening of the wrist extensor musculature
- Experimental (Experimental): Passive and active analytical stretching exercises described by Neiger and Simons , applying them to the muscle chain involved in lateral epicondylitis described by Busquet
  Interventions: Other: Passive and active analytical stretching exercises

INTERVENTIONS:
Other: Passive and active analytical stretching exercises — For each stretching technique described, 3 repetitions of 15 seconds duration will be performed of 15 seconds duration each, within the patient's tolerance threshold. In any case, the impossibility of performing any technique due to exacerbation of pain shall be recorded in a patient record created for this study, noting the technique in question and the reason for its technique in question and the reason for its non-application. Passive stretches shall be applied in the same order for all subjects.
  The physiotherapists in charge of applying the treatments will be trained in advance in the different techniques to be applied and will not in the different techniques to be applied and shall not intervene at any time in the two previous phases.
  Both the control group and the study group will receive their respective treatments two days a week for four weeks. In no case will any other type of treatment be associated treatment during the whole process.
  Arms: Experimental
Other: Static stretching of the extensor carpi radialis brevis and eccentric strengthening of the wrist extensor musculature — Static stretching of the extensor carpi radialis brevis and eccentric strengthening of the wrist extensor musculature
  Arms: Control group

SUMMARY:
Evaluation of the applying a stretching protocol to lateral epicondylitis.

DETAILED DESCRIPTION:
Epicondylitis is one of the most common soft tissue disorders of the locomotor system of the upper limb. Despite the existence of a large number of therapeutic alternatives for this type of injury, no agreed treatment protocol has been found. Some authors even suggest treating the patient from a more global biomechanical perspective.

OBJECTIVES. To evaluate the efficacy of applying a stretching protocol to the entire muscle chain involved in this injury and circumscribed to the entire affected upper limb.

METHODOLOGY. The study will be made up of 40 patients of both genders, randomly distributed in two groups: a control group made up of twenty patients to whom the usual Physiotherapy treatment will be applied, and an experimental group made up of the rest of the subjects, in which a stretching protocol will be applied to the whole upper limb affected and defined for this study. The evaluation process will consist of measuring pain perception using a visual analogue scale (VAS) and grip strength with a dynamometer. These measurements will be performed on all study subjects before starting treatment, at week 4 and week 6.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects over 18 years of age.
* Clinical diagnosis of lateral epicondylitis made by the Rehabilitation Physicians collaborating in this study.
* Patient's prior informed consent for inclusion in the study.

Exclusion Criteria:

* Patients with significant psychological, neurological and physical impairments that would prevent the recruitment of the information necessary for the research.
* Patients with significant psychological, neurological and physical alterations that would prevent the application of the treatments necessary for the research.
* Patients in a situation of legal litigation that could be affected by their participation in this study.
* Refusal to participate in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-30 (Estimated); Primary Completion 2022-05-03 (Estimated); Study Completion 2023-05-05 (Estimated)

PRIMARY OUTCOMES:
Elbow Pain | 1,5 months
  Measurement of pain perception: by means of a visual analogue scale (VAS), consisting of drawing a 100 mm long line in a centred position on a DINA A4 paper, cut with a segment perpendicular to it at each end. After informing the subject that the left and right segments represent the absence of pain and the maximum pain imaginable respectively, the subject is asked to point with a pencil on the line to the point where their pain is located.
Grip strength | 1,5 months
  A dynamometer shall be used for the test. Special care was taken to ensure that all subjects had the same position in order to be able to compare results. After informing the patient how to perform this test, the evaluation process consists of performing a maximum grip force for three seconds, executing it three times and with a minimum time interval of 60 seconds between them to avoid muscle fatigue. After completion of the test, the arithmetic mean of the results will be considered as the result.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Martin, Study Director — Cadiz University

IPD SHARING:
Plan to Share IPD: Yes
Publication in journals indexed in the Journal Citation Report (JCR),in the field of Rehabilitation and Physical Medicine and Physiotherapy.
  2. Dissemination of results in national and international Congresses of Rehabilitation and Physical Medicine and Physiotherapy.
  3. Dissemination to the public, press releases and explanatory brochures of the project.
Supporting Information: Study Protocol
Time Frame: In two years. In December 2023.
Access Criteria: open file

REFERENCES:
- [Background] Knutsen EJ, Calfee RP, Chen RE, Goldfarb CA, Park KW, Osei DA. Factors associated with failure of nonoperative treatment in lateral epicondylitis. Am J Sports Med. 2015 Sep;43(9):2133-7. doi: 10.1177/0363546515590220. Epub 2015 Jun 29. PMID 26122386
- [Background] Sanders TL Jr, Maradit Kremers H, Bryan AJ, Ransom JE, Smith J, Morrey BF. The epidemiology and health care burden of tennis elbow: a population-based study. Am J Sports Med. 2015 May;43(5):1066-71. doi: 10.1177/0363546514568087. Epub 2015 Feb 5. PMID 25656546
- [Background] Haahr JP, Andersen JH. Physical and psychosocial risk factors for lateral epicondylitis: a population based case-referent study. Occup Environ Med. 2003 May;60(5):322-9. doi: 10.1136/oem.60.5.322. PMID 12709516
- [Background] Fathy AA. Iontophoresis Versus Cyriax-Type exercises in Chronic Tennis Elbow among industrial workers. Electron Physician. 2015 Sep 16;7(5):1277-83. doi: 10.14661/1277. eCollection 2015 Sep. PMID 26435828
- [Background] Shiri R, Viikari-Juntura E, Varonen H, Heliovaara M. Prevalence and determinants of lateral and medial epicondylitis: a population study. Am J Epidemiol. 2006 Dec 1;164(11):1065-74. doi: 10.1093/aje/kwj325. Epub 2006 Sep 12. PMID 16968862
- [Background] Greenbaum B, Itamura J, Vangsness CT, Tibone J, Atkinson R. Extensor carpi radialis brevis. An anatomical analysis of its origin. J Bone Joint Surg Br. 1999 Sep;81(5):926-9. doi: 10.1302/0301-620x.81b5.9566. PMID 10530864
- [Background] Coel M, Yamada CY, Ko J. MR imaging of patients with lateral epicondylitis of the elbow (tennis elbow): importance of increased signal of the anconeus muscle. AJR Am J Roentgenol. 1993 Nov;161(5):1019-21. doi: 10.2214/ajr.161.5.8273602.
- [Background] Baker CL Jr, Murphy KP, Gottlob CA, Curd DT. Arthroscopic classification and treatment of lateral epicondylitis: two-year clinical results. J Shoulder Elbow Surg. 2000 Nov-Dec;9(6):475-82. doi: 10.1067/mse.2000.108533. PMID 11155299
- [Background] Babaei-Ghazani A, Shahrami B, Fallah E, Ahadi T, Forough B, Ebadi S. Continuous shortwave diathermy with exercise reduces pain and improves function in Lateral Epicondylitis more than sham diathermy: A randomized controlled trial. J Bodyw Mov Ther. 2020 Jan;24(1):69-76. doi: 10.1016/j.jbmt.2019.05.025. Epub 2019 May 24. PMID 31987565
- [Background] Yelland M, Rabago D, Ryan M, Ng SK, Vithanachchi D, Manickaraj N, Bisset L. Prolotherapy injections and physiotherapy used singly and in combination for lateral epicondylalgia: a single-blinded randomised clinical trial. BMC Musculoskelet Disord. 2019 Nov 3;20(1):509. doi: 10.1186/s12891-019-2905-5. PMID 31679521
- [Background] Reyhan AC, Sindel D, Dereli EE. The effects of Mulligan's mobilization with movement technique in patients with lateral epicondylitis. J Back Musculoskelet Rehabil. 2020;33(1):99-107. doi: 10.3233/BMR-181135. PMID 31104005
- [Background] Buchbinder R, Green SE, Struijs P. Tennis elbow. BMJ Clin Evid. 2008 May 28;2008:1117. PMID 19450309
- [Background] Nirschl RP. Elbow tendinosis/tennis elbow. Clin Sports Med. 1992 Oct;11(4):851-70. PMID 1423702
- [Background] Terra BB, Rodrigues LM, Filho AN, de Almeida GD, Cavatte JM, De Nadai A. Arthroscopic treatment for chronic lateral epicondylitis. Rev Bras Ortop. 2015 Jul 9;50(4):395-402. doi: 10.1016/j.rboe.2015.06.015. eCollection 2015 Jul-Aug. PMID 26401498
- [Background] Seng C, Mohan PC, Koh SB, Howe TS, Lim YG, Lee BP, Morrey BF. Ultrasonic Percutaneous Tenotomy for Recalcitrant Lateral Elbow Tendinopathy: Sustainability and Sonographic Progression at 3 Years. Am J Sports Med. 2016 Feb;44(2):504-10. doi: 10.1177/0363546515612758. Epub 2015 Nov 24. PMID 26602153
- [Background] Abbott JH. Mobilization with movement applied to the elbow affects shoulder range of movement in subjects with lateral epicondylalgia. Man Ther. 2001 Aug;6(3):170-7. doi: 10.1054/math.2001.0407. PMID 11527457
- [Background] Lucado AM, Kolber MJ, Cheng MS, Echternach JL Sr. Upper extremity strength characteristics in female recreational tennis players with and without lateral epicondylalgia. J Orthop Sports Phys Ther. 2012 Dec;42(12):1025-31. doi: 10.2519/jospt.2012.4095. Epub 2012 Sep 5. PMID 22960729
- [Background] Madding SW, Wong JG, Hallum A, Medeiros J. Effect of duration of passive stretch on hip abduction range of motion. J Orthop Sports Phys Ther. 1987;8(8):409-16. doi: 10.2519/jospt.1987.8.8.409. PMID 18797037
- [Background] Romero-Dapueto C, Mahn J, Cavada G, Daza R, Ulloa V, Antunez M. [Hand grip strength values in normal Chilean subjects]. Rev Med Chil. 2019 Jun;147(6):741-750. doi: 10.4067/S0034-98872019000600741. Spanish. PMID 31859827
- [Background] Viswas R, Ramachandran R, Korde Anantkumar P. Comparison of effectiveness of supervised exercise program and Cyriax physiotherapy in patients with tennis elbow (lateral epicondylitis): a randomized clinical trial. ScientificWorldJournal. 2012;2012:939645. doi: 10.1100/2012/939645. Epub 2012 May 2. PMID 22629225